CLINICAL TRIAL: NCT06243900
Title: NIRS: a Tool for the Diagnosis of Residual Renal Function Injury in Hemodialysis Patients
Brief Title: NIRS for the Diagnosis of Residual Renal Function Injury in Hemodialysis Patients
Acronym: HDRRFI-NIRS
Status: Enrolling by invitation | Type: Observational
Sponsor: Yuanjun Yang (Other)
Responsible Party: Sponsor-Investigator, Yuanjun Yang, Director, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: S2023-439-01
Record Dates: First submitted 2024-01-23; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: End-stage Renal Disease (ESRD)
Keywords: Hemodialysis; residual renal function; near-infrared spectroscopy
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The peripheral blood samples are mainly used to detect creatinine, urea, hemoglobin, C-reactive protein (CRP), IL-6, etc. The urine samples are mainly used to detect kidney injury markers, such as TFF3, KIM-1, IP-10, etc.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hemodialysis (HD) is the main renal replacement therapy for patients with end-stage renal disease (ESRD), accounting for approximately 69% of all renal replacement therapies and 89% of all dialysis. However, factors such as unstable hemodynamics have led to the gradual loss of residual renal function (RRF) in HD patients, which not only affects the adequacy of dialysis and complications control but also impacts their quality of life and survival. Unfortunately, until now, there have been no effective methods for early diagnosis and prediction of residual renal injury, and by the time it was discovered, the opportunity for effective treatment had been missed. The purpose of this study is to validate the value of near-infrared spectroscopy (NIRS) in the early diagnosis and prediction of residual renal injury. This will provide a basis for the application of NIRS in the early monitoring of residual renal injury in HD patients and offer a new method and perspective for the early diagnosis of residual renal injury in HD patients.

DETAILED DESCRIPTION:
Hemodialysis (HD) is the main renal replacement therapy for patients with end-stage renal disease (ESRD), accounting for approximately 69% of all renal replacement therapies and 89% of all dialysis. However, factors such as unstable hemodynamics have led to the gradual loss of residual renal function (RRF) in HD patients. Research has found that 25%-67% of HD patients progress to anuria within the first 10 months of starting dialysis. The rate of loss is much faster than peritoneal dialysis（PD）, and the more frequent the dialysis sessions, the faster the loss of RRF. The loss of RRF not only affects the adequacy of dialysis and complications control but also impacts the patient's quality of life and survival. Unfortunately, until now, there have been no effective methods for early diagnosis and prediction of residual renal injury.

Traditionally, monitoring and diagnosing kidney damage have relied mainly on serum creatinine, urine output, and estimated glomerular filtration rate (eGFR). However, these indicators often occur after kidney damage has occurred, and their detection is delayed. The sensitivity for early diagnosis of kidney injury is low. By the time abnormalities are detected, the crucial treatment opportunity may have been missed. In addition, serum creatinine and other tests are susceptible to factors such as fluid dilution and reduced production in the body. Although some biomarkers for early diagnosis of acute kidney injury (AKI) have been developed domestically and internationally, most of them have not been applied in clinical practice and cannot be monitored in real-time. Moreover, these biomarkers may have significant differences in their generation between AKI and end-stage renal disease (ESRD) patients, making them unsuitable for early diagnosis and monitoring of residual renal injury in HD patients.

Near-infrared spectroscopy (NIRS) is a simple, safe, non-invasive, and real-time detection method that reflects organ perfusion by measuring changes in regional oxygen saturation. It is widely used in the diagnosis and prediction of neurological disorders, early prediction of AKI related to surgical procedures (cardiovascular, digestive, neurological, etc.), and monitoring of renal perfusion function after kidney transplantation. In theory, it can also be used for early diagnosis of residual renal injury in HD patients. This study is an exploratory research aiming to validate the value of NIRS in early diagnosis of residual renal injury by analyzing the correlation between renal oxygen saturation and urine output, as well as eGFR.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Clinical diagnosis of end-stage renal disease requiring long-term hemodialysis treatment, with dialysis duration ≤ 3 months;
* Urine output > 500ml/day or GFR > 3ml/min/1.72m2;
* Signed and dated informed consented is obtained.

Exclusion Criteria:

* Presence of vascular access dysfunction (blood flow rate < 180ml/min);
* COPD or blood oxygen saturation < 95%;
* Severe heart failure;
* Active infection;
* Infectious disease;
* Distance between the kidney and body surface > 4cm;
* Severe pigmentation or skin lesions in the renal area;
* Patients with severe anemia;
* Patients with polycystic kidney disease;
* Expected dialysis duration < 6 months;
* Pregnancy or lactation women;
* Patients who are participating in other clinical studies, or who have participated in other clinical studies within 3 months prior to enrollment;
* Unwillingness to be followed up or poor adherence to treatment;
* Other circumstances that the investigator considers unsuitable for enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical diagnosis of end-stage renal disease requiring long-term hemodialysis treatment, with dialysis duration ≤ 3 months;
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-02-14 (Estimated)

PRIMARY OUTCOMES:
Change in the renal cerebral oxygen saturation | 10 months
  Measured by Near Infrared Spectroscopy
time to anuria | 10 months
  defined as ≤100 ml/d or ≤200 ml of urine volume in the short interdialytic period
residual renal function (RRF) | 10 months
  The RRF was calculated from an interdialytic urine collection and pre- and post-dialysate blood samples as the mean of the urea and creatinine clearances adjusted for body surface area using a "GFR calculator"

SECONDARY OUTCOMES:
serum creatinine | 10 months
  Taking a blood test to evaluation creatinine
serum urea nitrogen | 10 months
  Taking a blood test to evaluation urea nitrogen
C-reactive protein (CRP) | 10 months
  Taking a blood test to evaluation CRP
Interleukin-6 | 10 months
  Taking a blood test to evaluation Interleukin-6
TFF3 | 10 months
  Taking a urine test to evaluation TFF3
KIM-1 | 10 months
  Taking a urine test to evaluation KIM-1
IP-10 | 10 months
  Taking a urine test to evaluation IP-10

OTHER OUTCOMES:
hemoglobin | 10 months
  Collect data at baseline and during each follow-up visit.
systolic pressure | 10 months
  Collect data at baseline and during each follow-up visit.
diastolic pressure | 10 months
  Collect data at baseline and during each follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Guangyan Cai, PhD, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Koyner JL, Vaidya VS, Bennett MR, Ma Q, Worcester E, Akhter SA, Raman J, Jeevanandam V, O'Connor MF, Devarajan P, Bonventre JV, Murray PT. Urinary biomarkers in the clinical prognosis and early detection of acute kidney injury. Clin J Am Soc Nephrol. 2010 Dec;5(12):2154-65. doi: 10.2215/CJN.00740110. Epub 2010 Aug 26. PMID 20798258
- [Background] Hayek SS, Landsittel DP, Wei C, Zeier M, Yu ASL, Torres VE, Roth S, Pao CS, Reiser J. Soluble Urokinase Plasminogen Activator Receptor and Decline in Kidney Function in Autosomal Dominant Polycystic Kidney Disease. J Am Soc Nephrol. 2019 Jul;30(7):1305-1313. doi: 10.1681/ASN.2018121227. Epub 2019 Jun 6. PMID 31171572
- [Background] Bello AK, Okpechi IG, Osman MA, Cho Y, Htay H, Jha V, Wainstein M, Johnson DW. Epidemiology of haemodialysis outcomes. Nat Rev Nephrol. 2022 Jun;18(6):378-395. doi: 10.1038/s41581-022-00542-7. Epub 2022 Feb 22. PMID 35194215
- [Background] Ogata K. Clinicopathological study of kidneys from patients on chronic dialysis. Kidney Int. 1990 May;37(5):1333-40. doi: 10.1038/ki.1990.119. PMID 2345429
- [Background] Rottembourg J. Residual renal function and recovery of renal function in patients treated by CAPD. Kidney Int Suppl. 1993 Feb;40:S106-10. No abstract available. PMID 8445831
- [Background] Moist LM, Port FK, Orzol SM, Young EW, Ostbye T, Wolfe RA, Hulbert-Shearon T, Jones CA, Bloembergen WE. Predictors of loss of residual renal function among new dialysis patients. J Am Soc Nephrol. 2000 Mar;11(3):556-564. doi: 10.1681/ASN.V113556. PMID 10703680
- [Background] Misra M, Vonesh E, Van Stone JC, Moore HL, Prowant B, Nolph KD. Effect of cause and time of dropout on the residual GFR: a comparative analysis of the decline of GFR on dialysis. Kidney Int. 2001 Feb;59(2):754-63. doi: 10.1046/j.1523-1755.2001.059002754.x. PMID 11168959
- [Background] Jansen MA, Hart AA, Korevaar JC, Dekker FW, Boeschoten EW, Krediet RT; NECOSAD Study Group. Predictors of the rate of decline of residual renal function in incident dialysis patients. Kidney Int. 2002 Sep;62(3):1046-53. doi: 10.1046/j.1523-1755.2002.00505.x. PMID 12164889
- [Background] Teruel-Briones JL, Fernandez-Lucas M, Rivera-Gorrin M, Ruiz-Roso G, Diaz-Dominguez M, Rodriguez-Mendiola N, Quereda-Rodriguez-Navarro C. Progression of residual renal function with an increase in dialysis: haemodialysis versus peritoneal dialysis. Nefrologia. 2013;33(5):640-9. doi: 10.3265/Nefrologia.pre2013.May.12038. English, Spanish. PMID 24089155
- [Background] Daugirdas JT, Greene T, Rocco MV, Kaysen GA, Depner TA, Levin NW, Chertow GM, Ornt DB, Raimann JG, Larive B, Kliger AS; FHN Trial Group. Effect of frequent hemodialysis on residual kidney function. Kidney Int. 2013 May;83(5):949-58. doi: 10.1038/ki.2012.457. Epub 2013 Jan 23. PMID 23344474
- [Background] Obi Y, Streja E, Rhee CM, Ravel V, Amin AN, Cupisti A, Chen J, Mathew AT, Kovesdy CP, Mehrotra R, Kalantar-Zadeh K. Incremental Hemodialysis, Residual Kidney Function, and Mortality Risk in Incident Dialysis Patients: A Cohort Study. Am J Kidney Dis. 2016 Aug;68(2):256-265. doi: 10.1053/j.ajkd.2016.01.008. Epub 2016 Feb 9. PMID 26867814
- [Background] Wong J, Vilar E, Davenport A, Farrington K. Incremental haemodialysis. Nephrol Dial Transplant. 2015 Oct;30(10):1639-48. doi: 10.1093/ndt/gfv231. Epub 2015 Jun 1. PMID 26038351
- [Background] Bargman JM, Golper TA. The importance of residual renal function for patients on dialysis. Nephrol Dial Transplant. 2005 Apr;20(4):671-3. doi: 10.1093/ndt/gfh723. Epub 2005 Mar 8. No abstract available. PMID 15755759
- [Background] Wang AY, Lai KN. The importance of residual renal function in dialysis patients. Kidney Int. 2006 May;69(10):1726-32. doi: 10.1038/sj.ki.5000382. PMID 16612329
- [Background] Bragg-Gresham JL, Fissell RB, Mason NA, Bailie GR, Gillespie BW, Wizemann V, Cruz JM, Akiba T, Kurokawa K, Ramirez S, Young EW. Diuretic use, residual renal function, and mortality among hemodialysis patients in the Dialysis Outcomes and Practice Pattern Study (DOPPS). Am J Kidney Dis. 2007 Mar;49(3):426-31. doi: 10.1053/j.ajkd.2006.12.012. PMID 17336704
- [Background] Suda T, Hiroshige K, Ohta T, Watanabe Y, Iwamoto M, Kanegae K, Ohtani A, Nakashima Y. The contribution of residual renal function to overall nutritional status in chronic haemodialysis patients. Nephrol Dial Transplant. 2000 Mar;15(3):396-401. doi: 10.1093/ndt/15.3.396. PMID 10692527
- [Background] Shemin D, Bostom AG, Laliberty P, Dworkin LD. Residual renal function and mortality risk in hemodialysis patients. Am J Kidney Dis. 2001 Jul;38(1):85-90. doi: 10.1053/ajkd.2001.25198. PMID 11431186
- [Background] Delrue C, De Bruyne S, Speeckaert MM. The Potential Use of Near- and Mid-Infrared Spectroscopy in Kidney Diseases. Int J Mol Sci. 2023 Apr 4;24(7):6740. doi: 10.3390/ijms24076740. PMID 37047712
- [Background] Sakaki K, Kitamura T, Kohira S, Torii S, Mishima T, Hanayama N, Kobayashi K, Ohkubo H, Miyaji K. Regional thigh tissue oxygen saturation during cardiopulmonary bypass predicts acute kidney injury after cardiac surgery. J Artif Organs. 2020 Dec;23(4):315-320. doi: 10.1007/s10047-020-01175-y. Epub 2020 May 24. PMID 32448955
- [Background] Yu Y, Wu H, Liu C, Zhang C, Song Y, Ma Y, Li H, Lou J, Liu Y, Cao J, Zhang H, Xu Z, Evans RG, Duan C, Mi W. Intraoperative renal desaturation and postoperative acute kidney injury in older patients undergoing liver resection: A prospective cohort study. J Clin Anesth. 2023 Aug;87:111084. doi: 10.1016/j.jclinane.2023.111084. Epub 2023 Mar 9. PMID 36905791